CLINICAL TRIAL: NCT03867032
Title: Auditory Training With Speech Related Acoustic Cues Using Psychophysical Testing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI passed away. Ending grant and closing down lab
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Heather Wright, Professor, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Zhou_R01_study5
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear implant users (Experimental): The group will receive auditory training (psychophysical), and will be evaluated for speech recognition to determine the effect of training.
  Interventions: Behavioral: Auditory training

INTERVENTIONS:
Behavioral: Auditory training — Training with psychophysical tests (amplitude modulation detection on single electrodes) for improving speech recognition

SUMMARY:
In this study, the investigators will evaluate whether auditory training with speech-related acoustic features in psychophysical testing will help CI subjects improve speech recognition. The primary endpoint is the speech recognition measures.

ELIGIBILITY:
Inclusion Criteria:

* Native speakers of English
* Cochlear Nucleus cochlear implant users or Advanced Bionics users
* Postlingually deafened
* Has had device experience for at least one year
* Can be child or adult at the time of enrollment

Exclusion Criteria:

* None

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2022-12-26 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
speech recognition after training | starting 12 months after the award and will take up to 3.5 years to complete
  Subjects will be measured for their baseline speech recognition performance (A) and then measured again for speech recognition after receiving auditory training using the psychophysical methods (B). Finally, the subjects will be measured for speech recognition the third time after the training is withdrawn following a ABA longitudinal design.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banai K, Hornickel J, Skoe E, Nicol T, Zecker S, Kraus N. Reading and subcortical auditory function. Cereb Cortex. 2009 Nov;19(11):2699-707. doi: 10.1093/cercor/bhp024. Epub 2009 Mar 17. PMID 19293398
- [Background] Baumann S, Joly O, Rees A, Petkov CI, Sun L, Thiele A, Griffiths TD. The topography of frequency and time representation in primate auditory cortices. Elife. 2015 Jan 15;4:e03256. doi: 10.7554/eLife.03256. PMID 25590651
- [Background] Boebinger D, Evans S, Rosen S, Lima CF, Manly T, Scott SK. Musicians and non-musicians are equally adept at perceiving masked speech. J Acoust Soc Am. 2015 Jan;137(1):378-87. doi: 10.1121/1.4904537. PMID 25618067
- [Background] Chen JK, Chuang AY, McMahon C, Hsieh JC, Tung TH, Li LP. Music training improves pitch perception in prelingually deafened children with cochlear implants. Pediatrics. 2010 Apr;125(4):e793-800. doi: 10.1542/peds.2008-3620. Epub 2010 Mar 8. PMID 20211951
- [Background] Coffey EBJ, Mogilever NB, Zatorre RJ. Speech-in-noise perception in musicians: A review. Hear Res. 2017 Sep;352:49-69. doi: 10.1016/j.heares.2017.02.006. Epub 2017 Feb 14. PMID 28213134
- [Background] Fritz J, Elhilali M, Shamma S. Active listening: task-dependent plasticity of spectrotemporal receptive fields in primary auditory cortex. Hear Res. 2005 Aug;206(1-2):159-76. doi: 10.1016/j.heares.2005.01.015. PMID 16081006
- [Background] Fitzgerald MB, Wright BA. Perceptual learning and generalization resulting from training on an auditory amplitude-modulation detection task. J Acoust Soc Am. 2011 Feb;129(2):898-906. doi: 10.1121/1.3531841. PMID 21361447
- [Background] Fu QJ, Galvin JJ 3rd, Wang X, Wu JL. Benefits of music training in mandarin-speaking pediatric cochlear implant users. J Speech Lang Hear Res. 2015 Feb;58(1):163-9. doi: 10.1044/2014_JSLHR-H-14-0127. PMID 25321148
- [Background] Huyck JJ, Wright BA. Learning, worsening, and generalization in response to auditory perceptual training during adolescence. J Acoust Soc Am. 2013 Aug;134(2):1172-82. doi: 10.1121/1.4812258. PMID 23927116
- [Background] Looi V, Gfeller K, Driscoll V. MUSIC APPRECIATION AND TRAINING FOR COCHLEAR IMPLANT RECIPIENTS: A REVIEW. Semin Hear. 2012 Nov 1;33(4):307-334. doi: 10.1055/s-0032-1329222. Epub 2012 Nov 19. PMID 23459244
- [Background] Parbery-Clark A, Skoe E, Kraus N. Musical experience limits the degradative effects of background noise on the neural processing of sound. J Neurosci. 2009 Nov 11;29(45):14100-7. doi: 10.1523/JNEUROSCI.3256-09.2009. PMID 19906958
- [Background] Patel AD. Why would Musical Training Benefit the Neural Encoding of Speech? The OPERA Hypothesis. Front Psychol. 2011 Jun 29;2:142. doi: 10.3389/fpsyg.2011.00142. eCollection 2011. PMID 21747773
- [Background] Polley DB, Steinberg EE, Merzenich MM. Perceptual learning directs auditory cortical map reorganization through top-down influences. J Neurosci. 2006 May 3;26(18):4970-82. doi: 10.1523/JNEUROSCI.3771-05.2006. PMID 16672673
- [Background] Ruggles DR, Freyman RL, Oxenham AJ. Influence of musical training on understanding voiced and whispered speech in noise. PLoS One. 2014 Jan 28;9(1):e86980. doi: 10.1371/journal.pone.0086980. eCollection 2014. PMID 24489819
- [Background] Sabin AT, Eddins DA, Wright BA. Perceptual learning evidence for tuning to spectrotemporal modulation in the human auditory system. J Neurosci. 2012 May 9;32(19):6542-9. doi: 10.1523/JNEUROSCI.5732-11.2012. PMID 22573676
- [Background] Szpiro SF, Wright BA, Carrasco M. Learning one task by interleaving practice with another task. Vision Res. 2014 Aug;101:118-24. doi: 10.1016/j.visres.2014.06.004. Epub 2014 Jun 21. PMID 24959653
- [Background] Wright BA, Sabin AT, Zhang Y, Marrone N, Fitzgerald MB. Enhancing perceptual learning by combining practice with periods of additional sensory stimulation. J Neurosci. 2010 Sep 22;30(38):12868-77. doi: 10.1523/JNEUROSCI.0487-10.2010. PMID 20861390
- [Background] Yucel E, Sennaroglu G, Belgin E. The family oriented musical training for children with cochlear implants: speech and musical perception results of two year follow-up. Int J Pediatr Otorhinolaryngol. 2009 Jul;73(7):1043-52. doi: 10.1016/j.ijporl.2009.04.009. Epub 2009 May 2. PMID 19411117